CLINICAL TRIAL: NCT00635245
Title: A Phase 1 Pharmacodynamic Study Of CP-751,871 As Neoadjuvant Treatment For Early Breast Cancer
Brief Title: CP-751871 In Treating Women With Early-Stage Breast Cancer That Can Be Removed By Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Masking: None | Purpose: Treatment
Other Study IDs: A4021012; P30CA077598 (NIH); NCI-CDR0000589252
Record Dates: First submitted 2008-03-12; First posted 2008-03-13 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — figitumumab; Magnetic Resonance Spectroscopy; Neoadjuvant Therapy

INTERVENTIONS:
Biological: figitumumab
Other: imaging biomarker analysis
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: conventional surgery
Procedure: magnetic resonance spectroscopic imaging
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as CP-751871, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase I trial is studying the side effects and best way to give CP-751871 in treating patients with early-stage breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
Primary

* To evaluate the change in total tumor choline levels in women with operable early breast cancer in response to neoadjuvant CP-751871 treatment.

Secondary

* To assess changes in tumor glucose levels after CP-751871 treatment using magnetic resonance spectroscopy in these patients.
* To assess the safety, tolerability, and immunogenicity of CP-751871 in these patients.
* To assess the effect of CP-751871 on Insulin-like Growth Factor 1 receptor (IGF-1R) signaling markers in tumor tissues in these patients.
* To assess the clinical efficacy of CP-751871 in these patients (MRI and pathological responses).

OUTLINE: Patients receive CP-751871 IV over 5 hours on days 1 and 22 and undergo magnetic resonance spectroscopy on days 8 and 29. Patients may also undergo surgery between days 29-43 to obtain a tumor sample for analysis of markers related to the IGR-1R pathway.

After completion of study treatment, patients will be followed for 5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed early operable adenocarcinoma of the breast
* No evidence of invasive lobular breast disease
* Measurable disease, defined as at least 1 lesion ≥ 2 cm by MRI
* Measurable levels of total choline according to institutional criteria by magnetic resonance spectroscopy
* Must have available or scheduled core breast biopsy procedure
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* Platelet count ≥ 100,000/mm^³
* Neutrophil count ≥ 1,500/mm³
* Creatinine < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* ALT and AST < 2.5 times ULN
* Fertile patients must use adequate barrier method contraception during and for at least 150 days after completion of study treatment
* Ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures
* No known hypersensitivity to monoclonal antibodies
* No prior or active malignancies other than curatively treated in situ carcinoma of the cervix, uterus, or basal cell or squamous cell carcinoma of the skin
* No serious uncontrolled medical disorder or active infection that would impair the ability to receive study treatment
* No significant active cardiac disease including any of the following:

  * Uncontrolled high blood pressure (i.e., systolic blood pressure [BP] > 160 mm Hg and diastolic BP > 95 mm Hg)
  * Unstable angina
  * Deep venous thrombosis
  * Pulmonary embolism
  * Cerebrovascular attack
  * Valvular disease
  * Congestive heart failure
  * Myocardial infarction with the past 6 months
  * Serious cardiac arrhythmias
* No dementia or significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with study requirements

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior surgery and recovered
* More than 2 weeks since high-dose corticosteroid therapy (i.e., ≥ 100 mg prednisone per day or > 40 mg dexamethasone per day)
* No prior anti-IGF-1R based investigational therapy
* No prior systemic therapy for primary disease
* No concurrent chronic systemic high-dose immunosuppressive steroid therapy

  * Low-dose steroids for nausea and vomiting control allowed
  * Topical corticosteroid applications, inhaled sprays, eye drops or local injections (e.g., intraocular) allowed
* No concurrent other anticancer drugs or therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Tumor total choline (tCho) changes determined by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Safety, tolerability and human anti-human antibodies (HAHA) response
Tissue markers
Measure of tumor glucose levels
Pathological response
Tumor size by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Yee, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota